CLINICAL TRIAL: NCT01614171
Title: Trial of Growth Hormone for Osteoporosis Pseudoglioma Syndrome
Brief Title: Growth Hormone for Osteoporosis Pseudoglioma Syndrome
Acronym: GHOPPG
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: it was never started because it was never funded
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Elizabeth Streeten, Associate Professor of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00053014
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2017-04

CONDITIONS: Osteoporosis Pseudoglioma Syndrome
Keywords: osteoporosis pseudoglioma; OPPG; growth hormone; osteoporosis
MeSH Terms: conditions — Exudative Vitreoretinopathy 4; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Growth hormone therapy (Experimental): Growth hormone treatment for 6 months
  Interventions: Biological: Human recombinant growth hormone

INTERVENTIONS:
Biological: Human recombinant growth hormone — growth hormone treatment for 6 months (daily, weight based)

SUMMARY:
Osteoporosis pseudoglioma (OPPG) syndrome is a rare autosomal recessive condition of childhood osteoporosis and congenital blindness for which new treatments are needed. We have found that body fat is increased in OPPG and muscle mass is reduced. We hypothesize that growth hormone therapy will improve muscle mass and bone strength in OPPG.

DETAILED DESCRIPTION:
Osteoporosis pseudoglioma (OPPG) syndrome is a rare autosomal recessive condition of childhood osteoporosis and congenital blindness for which new treatments are needed. We have found that body fat is increased in OPPG and muscle mass is reduced. We hypothesize that growth hormone therapy will improve muscle mass and bone strength in OPPG.

ELIGIBILITY:
Inclusion Criteria:

* Osteoporosis pseudoglioma syndrome
* Age 4 years and above
* not on medication for osteoporosis

Exclusion Criteria:

* pregnant
* Age under 4 yrs
* Active malignancy

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Bone quality by pQCT | 6 months
  By pQCT: periosteal circumference, cortical density, trabecular density, section modulus

SECONDARY OUTCOMES:
Body fat percent | 6 months
  Percent body fat by DXA

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Streeten, MD, Principal Investigator — University of Maryland School of Medicine, Division of Endocrinology
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States